CLINICAL TRIAL: NCT01590498
Title: Salvage Radiotherapy vs Observation for Castration Resistant Prostate Cancer in Central China
Brief Title: Radiotherapy vs Observation for CRPC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhengzhou University (Other)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other); the cancer hospital of Zhengzhou University (Unknown); People's Hospital of Zhengzhou University (Other); Xinyang Central Hospital (Other); Zhoukou Central Hospital (Other); the second people's hospital of kaifeng (Unknown)
Responsible Party: Principal Investigator, Liu Bingqian, Principal Investigator, Zhengzhou University
Other Study IDs: PCA0608; NNSFC (Other Grant/Funding Number: 30801151)
Record Dates: First submitted 2012-04-27; First posted 2012-05-03 (Estimated); Last update posted 2012-05-04 (Estimated); Status verified 2012-05

CONDITIONS: Hormone Refractory Prostate Cancer
Keywords: Adenocarcinoma; Prostatic Neoplasms; Carcinoma; Prostatic Diseases
MeSH Terms: conditions — Adenocarcinoma; Prostatic Neoplasms; Carcinoma; Prostatic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — the biopsy specimens of prostate tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Salvage radiotherapy: local radiation to the prostate and metastasis following biochemical or clinical recurrence
- observation: did not receive salvage following biochemical or clinical recurrence

SUMMARY:
The purpose of the study is to determine whether radiotherapy improves cancer control and overall survival among patients with Castration resistant prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Eligible patients had histologically or cytologically confirmed adenocarcinoma of the prostate with clinical or radiologic evidence of disease progression during hormonal therapy
2. Patients were receiving primary androgen-ablation therapy as maintenance therapy. At least four weeks had to have elapsed between the withdrawal of antiandrogens (six weeks in the case of bicalutamide) and enroll ment, so as to avoid the possibility of confounding as a result of the response to antiandrogen withdrawal.
3. Another requirement was disease progression, as indicated by increasing serum levels of PSA on three consecutive measurements obtained at least one week apart or findings on physical examination or imaging studies.
4. Normal cardiac function was required.

Exclusion Criteria:

1. patients had a Karnofsky performance-status score of at most 60 percent
2. prior treatment with cytotoxic agents or radioisotopes
3. with history of another cancer within the preceding five years, brain or leptomeningeal metastases, symptomatic peripheral neuropathy of grade 2 or higher, and other serious medical condition.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: inpatients with CRPC in 9 hospitals
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2012-05; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
overall survival | From the date of biochemical or clinical recurrence of prostate cancer following hormonal therapy to December 31, 2016 or date of death from any cause, whichever came first, assessed up to 3 years.

SECONDARY OUTCOMES:
prostate cancer specific mortality | From the date of biochemical or clinical recurrence of prostate cancer following hormonal therapy to December 31, 2016 or death from prostate cancer or treatment complications, whichever came first, assessed up to 3 years.

CONTACTS AND LOCATIONS:
Overall Officials: Liu Bingqian, MD Ph.D, Principal Investigator — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- the first affiliated hospital of Zhengzhou University, Zhengzhou, Henan, China